CLINICAL TRIAL: NCT04207307
Title: Best Function of Range of Motion (cRCT)
Acronym: bestform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Prof. Otto Beisheim Foundation (Other); Institute for Medical Informatics, Statistics and Epidemiology (IMedIS) (Unknown); Münchner Studienzentrum (MSZ) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bestform_122019
Record Dates: First submitted 2019-12-16; First posted 2019-12-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Mobility
Keywords: older people; oldest old; frailty; sarcopenia; exercise; resistance training; elderly; falls
MeSH Terms: conditions — Frailty; Sarcopenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial (1:1)
Who Masked: Outcomes Assessor
Masking Description: Primary endpoint is assessed by a rater who is otherwise not involved in the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal exercise intervention (Experimental): Behavioral: Multimodal exercise intervention with machine-based resistance, coordination and endurance training, 1-2 times per week for 30-45 min (increasing amount of training).
  Interventions: Behavioral: Multimodal exercise program
- Usual Care (Sham Comparator): General recommendations for healthy ageing, usual physical activity. No machine-based strength training intervention.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Multimodal exercise program — Multimodal exercise intervention (machine-based resistance, coordination and endurance training).
  Arms: Multimodal exercise intervention
Behavioral: Usual Care — General recommendations for healthy ageing, no machine-based strength training intervention.
  Arms: Usual Care

SUMMARY:
Mobility is a crucial factor for independence and quality of life in older people. However, the majority of those in retirement homes are not physically active to maintain mobility and independence.

The aim of the cluster randomized controlled bestform trial in 20 retirement homes (1:1 randomization) is to evaluate the efficacy of a multimodal exercise program for older people living in retirement homes in comparison to usual care over 6 months.

Within the intervention facilities, the participants will take part in a physical activity program over 6 months (2 times a week à 45 min) consisting of machine-based strength, coordination and endurance training.

Criteria of effectiveness are changes in physical function (primary endpoint: Change of Short Physical Performance Battery Score after 6 months) and the following secondary endpoints: mobility and balance, rate of falls, cardiometabolic risk factors, myocard function, quality of life and lifestyle factors (nutrition, physical activity), assessed by medical assessments, physical performance tests and various questionnaires after 3 and 6 months. Follow-up data will be collected after 18 and 30 months (questionnaire).

DETAILED DESCRIPTION:
Mobility is a crucial factor for independence and quality of life at old age. Particularly those in retirement homes have a reduced physical activity status.

The aim of the bestform trial is the integration of an exercise concept comprising resistance, coordination and endurance training in retirement homes to promote mobility and independence as well as to reduce the risk of falling in older people.

The study is organized and conducted as a multi-center, two-armed cluster randomized study in 20 retirement homes (1:1 randomization in intervention retirement homes and control retirement homes with usual care) in the area of Munich, Germany. A total of at least 400 older people will subsequently be recruited. It is expected to recruit n≥20 older people per participating retirement home.

The intervention group will participate in an exercise training for 6 months, which will take place in the period from March 2020 to October 2021 (extended until August 2023). The multimodal intervention consists of a machine-based resistance, coordination and endurance training, which is performed 1-2 times per week for 30-45 minutes with increasing amount of training. Age and disability adapted pneumatic resistance training machines are used targeting large muscle groups. The endurance training is performed on upright-bicycle and recumbent bicycle ergometers. Coordination is exercised statically on the floor or a balance pad and dynamically on a balance-platform according to the individual training plan.

The aim of the bestform trial is to examine the efficacy of this multimodal training on physical function measured by the Short Physical Performance Battery (SPPB) (primary endpoint) over a 6-month period.

In addition, the impact of the training on mobility and balance, physical capacity (6-min-walk test), rate of falls, anthropometric parameters, cardiometabolic risk parameters (echocardiography, blood parameters), fear of falling, quality of life and other life style factors (nutrition, physical activity) assessed by medical assessments, physical performance tests and various questionnaires will be investigated after 3 and 6 months. Follow-up data will be collected after 18 and 30 months (questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be resident of one of the participating retirement homes
* Written informed consent of the study participant or legal representative
* Being able to stand independently (without assistance)

Exclusion Criteria:

Any acute or chronic illness or physical/mental condition as well as any form of dementia, which does not allow to stand independently or which does not allow physical training in small groups or which would require a training with medical supervision

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 404 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Change in Short Physical Performance Battery | Baseline to 6 months
  The Short Physical Performance Battery is a summary performance score out of 3 tests (standing balance test, gait speed test, and chair-stand-test). Categories of performance will be formed for each performance test (0 points to 4 points) and a summary score will be used. The sum score ranges from 0 (worst performance) to 12 (best performance).

SECONDARY OUTCOMES:
Change in balance ability and mobility | Change after 3 and 6 months
  Change in balance ability and mobility is measured by the Timed-Up-and-Go-Test. A higher time needed (measured in seconds) in the test is associated with more deficits in mobility.
Change in physical capacity | Change after 3 and 6 months
  Change in physical capacity is measured by the 6-min-walk test. A lower distance (measured in meters) in the 6-min-walk test is associated with lower exercise capacity and general health status.
Change in handgrip strength | Change after 3 and 6 months
  Change in handgrip strength is measured by a hand dynamometer.
Rate of falls | 6 months
  Rate of falls is measured by a fall diary.
Change in body composition | Change after 3 and 6 months
  Change in body composition is measured by bioelectrical impedance analysis.
Change in body weight | Change after 3 and 6 months
  Change in body weight is measured with a scale. Weight and weight change in kilograms can be used to identify participants, who are at risk of obesity or malnutrition.
Change in calf circumference | Change after 3 and 6 months
  Change in calf circumference is measured by tape.
Change in cardiac function | Change after 6 months
  Change in cardiac function is measured by echocardiography.
Change in inflammatory marker | Change after 3 and 6 months
  Change in biomarkers associated with inflammation and immunological function.
Change in brain-derived neutrophic factor | Change after 3 and 6 months
  Change in brain-derived neutrophic factor is measured by the concentration of brain-derived neutrophic factor in serum.
Change in fear of falling | Change after 3 and 6 months
  Change in fear of falling is measured by the short Falls Efficacy Scale questionnaire. The questionnaire comprises 7 items with 4 answer options (0 to 4 points). To obtain the total score, the sum of points of all answers was calculated. A higher score indicates a higher level of fear of falling.
Change in quality of life | Change after 3 and 6 months
  Change in quality of life is measured by WHO-5 (Well-Being Index) questionnaire. The questionnaire comprises 5 statements about the feeling over the past 2 weeks (0 to 5 points). The raw score is multiplied by 4. The final score range from 0 (worst imaginable well-being) to 100 (best imaginable well-being).
Change in nutritional status | Change after 3 and 6 months
  Change in nutritional status is measured by Mini Nutritional Assessment (MNA®-SF). The questionnaire comprises 6 questions. The sum of points of all answers is calculated. 12-14 points indicate a normal nutritional status, 8-11 points a risk of malnutrition, and 0-7 points is classified as malnourished.
Change in activity of daily living | Change after 3 and 6 months
  Change in activity of daily living is measured by the Barthel-Index. The Barthel-Index comprises 10 items (0-15 points). The sum of points of all answers is calculated. Lower scores indicate a higher grade of disability.
Change in risk for sarcopenia | Change after 3 and 6 months
  Change in risk for sarcopenia is measured by SARC-F-questionnaire. The questionnaire comprises five components. The sum of points of all answers is calculated. The sum score ranges from 0 (best) to 10 (worst).
Change in cognition | Change after 6 months
  Changes in cognition is measured by the Montreal Cognitive Assessment (MoCA). The MoCA test is scored out of 30 points.
Change in Short Physical Performance Battery | Baseline to 3 months
  The Short Physical Performance Battery is a summary performance score out of 3 tests (standing balance test, gait speed test, and chair-stand-test). Categories of performance will be formed for each performance test (0 points to 4 points) and a summary score will be used. The sum score ranges from 0 (worst performance) to 12 (best performance).
Follow-up evaluation of MACE | Changes over 18 and 30 months
  Major adverse cardiac events (MACE) and all-cause mortality will be documented during the follow-up. MACE are cardiovascular death, non-fatal stroke, and non-fatal myocardial infarction (3-point MACE).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Halle, MD, Study Director — Department of Prevention, Rehabilitation and Sports Medicine
Locations (1):
- Department of Prevention, Rehabilitation and Sports Medicine, Faculty of Medicine, Technichal University of Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siegrist M, Schaller N, Weiss M, Isaak J, Schmid V, Koppel E, Weichenberger M, Mende E, Haller B, Halle M. Study protocol of a cluster-randomised controlled trial assessing a multimodal machine-based exercise training programme in senior care facilities over 6 months - the bestform study (best function of range of motion). BMC Geriatr. 2023 Aug 22;23(1):505. doi: 10.1186/s12877-023-04176-7. PMID 37605110